CLINICAL TRIAL: NCT05850975
Title: Do Mind Ease Interventions Reduce Feelings of Acute Anxiety? A Randomised Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: University of Bonn (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, JanBrauner, medical doctor, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R82884/RE001; https://osf.io/36ukh (Registry Identifier: OSF)
Record Dates: First submitted 2023-04-29; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Anxiety
Keywords: anxiety; app; psychotherapy; mindfulness; acceptance and commitment therapy; cognitive behavioural therapy; randomised controlled trial; depression
MeSH Terms: conditions — Anxiety Disorders; Alzheimer Disease; Depression | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to an intervention or control condition.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants are not told whether they are in an intervention or control condition. The app is both the care provider and the outcomes assessor. The investigator will be blinded while analysing the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- mindful breathing (Experimental)
  Interventions: Other: intervention with this name in MindEase app
- deep breathing (Experimental)
  Interventions: Other: intervention with this name in MindEase app
- cognitive therapy (Experimental)
  Interventions: Other: intervention with this name in MindEase app
- dare response (Experimental)
  Interventions: Other: intervention with this name in MindEase app
- defusion (Experimental)
  Interventions: Other: intervention with this name in MindEase app
- in flow with fear (Experimental)
  Interventions: Other: intervention with this name in MindEase app
- gratitude practice (Experimental)
  Interventions: Other: intervention with this name in MindEase app
- guided mindfulness (Experimental)
  Interventions: Other: intervention with this name in MindEase app
- muscle relaxation (Experimental)
  Interventions: Other: intervention with this name in MindEase app
- reframe your fears (Experimental)
  Interventions: Other: intervention with this name in MindEase app
- calming visualization (Experimental)
  Interventions: Other: intervention with this name in MindEase app
- reflective writing (Experimental)
  Interventions: Other: intervention with this name in MindEase app
- reading about anxiety (Placebo Comparator)
  Interventions: Other: reading about anxiety
- do what you would usually do (No Intervention)

INTERVENTIONS:
Other: intervention with this name in MindEase app — MindEase is an app which provides interventions against anxiety. The interventions are based on mindfulness, acceptance and commitment therapy, and cognitive behavioural therapy.
  Arms: calming visualization; cognitive therapy; dare response; deep breathing; defusion; gratitude practice; guided mindfulness; in flow with fear; mindful breathing; muscle relaxation; reflective writing; reframe your fears
Other: reading about anxiety — Participants are given an educational text to read about anxiety.
  Arms: reading about anxiety

SUMMARY:
This study investigates the short-term effects of the MindEase app on anxiety levels.

DETAILED DESCRIPTION:
Anxiety is a common symptom in the world's population (Whiteford et al., 2013). It occurs as a symptom within other mental disorders and as a disorder in itself (American Psychiatric Association, 2013).

There are several ways of dealing with anxiety, from short guidance for coping on a symptom level to professional health. (Emmelkamp & Ehring, 2014). Many people suffering from anxiety below a threshold indicating need for professional therapy may profit from strategies to calm down. (Helmchen & Linden, 2000). Among the strategies that are effective, there are guided interventions that people can use via a web-based interface on a computer or smartphone (Taylor et al., 2021). While it is known for most interventions that they are helpful, it is often unclear if they work also in web-based environments (Baumel et al., 2020). This is because most research regarding the topic investigates the effectiveness of mental-health apps as a whole, while research of specific interventions is missing (Domhardt et al., 2019). However, to develop effective apps, it is crucial to identify which specific interventions are most efficient in a web-based setting. (Domhardt et al., 2019; Firth et al., 2017). Therefore we want to identify interventions working effectively in an online format.

Mind Ease is an app that offers different established interventions within one framework to their users when they feel anxious. This framework makes the different interventions comparable to each other. For this reason, we will test the interventions that are used in the Mind Ease-app.

In a first study we will correlate the Mind Ease 3-sliders-score with the state-trait- anxiety-Inventory (SAI). In a second study we will measure participants'; acute anxiety (with the 3-sliders- score) before and after they performed a 10 minutes web-based cognitive or mindfulness-associated intervention. We will compare the anticipated reduction in anxiety to the reduction measured in participants in a control group.

Prospectively registered here: https://osf.io/36ukh

ELIGIBILITY:
Inclusion Criteria:

* anxiety score is above cut-off

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6200 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
change in anxiety score | immediately before and immediately after the intervention
  sum of three slider questions on emotional state (3-sliders-score)

CONTACTS AND LOCATIONS:
Overall Officials: Jan M Brauner, MD, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymous participant data will be accessible to anyone upon request.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Immediately after publication. No end date.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Derived] Sandkuhler JF, Kahl F, Sadurska MZ, Brietbart P, Greenberg S, Brauner J. The Immediate Impact of App-Based Psychotherapeutic Exercises on Anxiety: An RCT. Depress Anxiety. 2025 Apr 2;2025:5586831. doi: 10.1155/da/5586831. eCollection 2025. PMID 40225732